CLINICAL TRIAL: NCT03240003
Title: A Novel Computer-Based Therapy for Social Anxiety
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: funding unavailable
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Franklin Schneier, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 7527 (SAD)
Record Dates: First submitted 2017-07-25; First posted 2017-08-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety; Social Anxiety Disorder; SAD
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GC-MRT (Experimental): Group 1 will receive a 4-week (8-sessions) course of standard GC-MRT
  Interventions: Behavioral: GC-MRT
- non-GC-MRT (Active Comparator): Group 2 will receive a 4-week (8-sessions) course of non-GC-MRT
  Interventions: Behavioral: Non-GC-MRT
- GC-MRT-modified (Experimental): Group 3 will receive a 4-week (8-sessions) course of modified GC-MRT.
  Interventions: Behavioral: modified GC-MRT

INTERVENTIONS:
Behavioral: GC-MRT — Group 1 will receive a 4-week (8-sessions) course of GC-MRT
  Arms: GC-MRT
Behavioral: modified GC-MRT — group 3 will receive a 4-week (8-sessions) course of GC-MRT, modified
  Arms: GC-MRT-modified
Behavioral: Non-GC-MRT — Group 2 will receive a 4-week (8-sessions) course of non-GC-MRT
  Arms: non-GC-MRT

SUMMARY:
The present study is a double blind trial that seeks to examine the feasibility, acceptability, efficacy, and mechanism of a recently developed eye-tracking-based therapy (GC-MRT) in individuals with social anxiety disorder (SAD)

DETAILED DESCRIPTION:
The present study is a double blind trial that seeks to examine the feasibility, acceptability, efficacy, and mechanism of a recently developed eye-tracking-based therapy (GC-MRT) in individuals with social anxiety disorder (SAD). The purpose of this study is to assess whether a brief computer-based research treatment, provided in 30 minutes sessions twice a week for 4 weeks, helps improve social anxiety symptoms, and by what mechanism. The study will also assess the effect of research treatments on brain activity using a scan called magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 60
* Current DSM-V primary diagnosis of SAD
* Score of at least 50 on the Liebowitz Social Anxiety Scale (Self-rated version)
* Fluent in English and willing and able to give informed written consent and participate responsibly in the protocol
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Present or past psychotic episode, psychotic disorder, schizophrenia, schizoaffective disorder, or bipolar disorder
* Current severe depression
* Suicidal ideation or behavior
* Current diagnosis of PTSD, obsessive-compulsive disorder, bipolar disorder, manic episode or tic disorder
* Current or past organic mental disorder, seizure disorder, epilepsy or brain injury
* Current unstable or untreated medical illness
* Severe alcohol use disorder, severe cannabis use disorder, and any severity of other substance use disorder (except nicotine use disorders allowed)
* Use of psychiatric medication in the past month other than a stable dose of selective serotonin reuptake inhibitors (SSRIs) for a least 3 months
* Any concurrent cognitive behavioral therapy; other psychotherapy that was initiated in the past 3 months
* Pregnancy, or plans to become pregnant during the period of the study - will be assessed by Urine β-HCG
* Contraindication to MRI scanning:
* Paramagnetic metallic implants or devices contraindicating magnetic resonance imaging or any other non-removable paramagnetic metal in the body (e.g. pacemaker, paramagnetic metallic prosthesis, surgical clips, shrapnel, necessity for constant medicinal patch, some tattoos)
* Being unable to tolerate the scanning procedures (i.e., severe obesity, claustrophobia)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale | 4 months
  Total score of the Liebowitz Social Anxiety Scale

SECONDARY OUTCOMES:
Social Phobia Inventory (SPIN) | 4 months
  The Social Phobia Inventory (abbreviated as SPIN) is a self-rated questionnaire that will be used to assess severity of social anxiety Disorder. 17 items related to social anxiety each rated on a score of 0 to 4, with a minimum total score of 0 (least social anxiety), and a maximum total score of 68 (most social anxiety).
Quality of Life Enjoyment & Satisfaction Questionnaire | 4 months
  Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LES-Q): self-rated assessment of quality of life. 16 items related to life quality, each rated on a score of 1 (very poor) to 5 (very good), with a minimum total score of 16, and a maximum total score of 80.
Revised Social Anhedonia Scale | 4 months
  40-item self-rated social anhedonia scale. Items are comprised of statements that participants agree or disagree with, by answering "yes"(1), or "no"(0), with some items reverse-coded. The minimum score is 0 (least social anhedonia); maximum score is 40 (most social anhedonia).
Snaith Hamilton Pleasure Scale | 4 months
  Snaith Hamilton Pleasure Scale (SHAPS). Fourteen-item self-rated anhedonia scale. Items were comprised of statements that participants rated as "strongly disagree" (1), "disagree" (2), "agree" (3), or "strongly agree" (4). The lowest possible score was 14, the highest possible score was 56 (greatest anhedonia)
Hamilton Rating Scale for Depression - 17 item version | 4 months
  Hamilton Rating Scale for Depression -17 item version. This standard scale will be used to assess severity of depression, minimum score is 0 (least depression); maximum score is 50 (greatest depression).
Clinical Global Impression-Change Scale | 4 months
  Clinical Global Impression-Change Scale: A quickly administered and widely used observer rating, with rating from 1 (very much improved) to 7 (very much worse). Responder category is defined by a score of 1 or 2.

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Schneier, MD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chevallier C, Tonge N, Safra L, Kahn D, Kohls G, Miller J, Schultz RT. Measuring Social Motivation Using Signal Detection and Reward Responsiveness. PLoS One. 2016 Dec 1;11(12):e0167024. doi: 10.1371/journal.pone.0167024. eCollection 2016. PMID 27907025
- [Background] Cisler JM, Koster EH. Mechanisms of attentional biases towards threat in anxiety disorders: An integrative review. Clin Psychol Rev. 2010 Mar;30(2):203-16. doi: 10.1016/j.cpr.2009.11.003. Epub 2009 Dec 14. PMID 20005616
- [Background] Gur RC, Schroeder L, Turner T, McGrath C, Chan RM, Turetsky BI, Alsop D, Maldjian J, Gur RE. Brain activation during facial emotion processing. Neuroimage. 2002 Jul;16(3 Pt 1):651-62. doi: 10.1006/nimg.2002.1097. PMID 12169250
- [Background] Heeren A, Mogoase C, Philippot P, McNally RJ. Attention bias modification for social anxiety: A systematic review and meta-analysis. Clin Psychol Rev. 2015 Aug;40:76-90. doi: 10.1016/j.cpr.2015.06.001. Epub 2015 Jun 6. PMID 26080314
- [Background] Klumpp H, Angstadt M, Phan KL. Shifting the focus of attention modulates amygdala and anterior cingulate cortex reactivity to emotional faces. Neurosci Lett. 2012 Apr 18;514(2):210-3. doi: 10.1016/j.neulet.2012.03.003. Epub 2012 Mar 8. PMID 22425719
- [Background] Klumpp H, Post D, Angstadt M, Fitzgerald DA, Phan KL. Anterior cingulate cortex and insula response during indirect and direct processing of emotional faces in generalized social anxiety disorder. Biol Mood Anxiety Disord. 2013 Apr 2;3:7. doi: 10.1186/2045-5380-3-7. eCollection 2013. PMID 23547713
- [Background] Lazarov A, Abend R, Bar-Haim Y. Social anxiety is related to increased dwell time on socially threatening faces. J Affect Disord. 2016 Mar 15;193:282-8. doi: 10.1016/j.jad.2016.01.007. Epub 2016 Jan 12. PMID 26774515
- [Background] Lazarov A, Pine DS, Bar-Haim Y. Gaze-Contingent Music Reward Therapy for Social Anxiety Disorder: A Randomized Controlled Trial. Am J Psychiatry. 2017 Jul 1;174(7):649-656. doi: 10.1176/appi.ajp.2016.16080894. Epub 2017 Jan 20. PMID 28103714
- [Background] Linetzky M, Pergamin-Hight L, Pine DS, Bar-Haim Y. Quantitative evaluation of the clinical efficacy of attention bias modification treatment for anxiety disorders. Depress Anxiety. 2015 Jun;32(6):383-91. doi: 10.1002/da.22344. Epub 2015 Feb 24. PMID 25708991
- [Background] Mogoase C, David D, Koster EH. Clinical efficacy of attentional bias modification procedures: an updated meta-analysis. J Clin Psychol. 2014 Dec;70(12):1133-57. doi: 10.1002/jclp.22081. Epub 2014 Mar 20. PMID 24652823
- [Background] Morrison AS, Heimberg RG. Social anxiety and social anxiety disorder. Annu Rev Clin Psychol. 2013;9:249-74. doi: 10.1146/annurev-clinpsy-050212-185631. PMID 23537485
- [Background] Richey JA, Rittenberg A, Hughes L, Damiano CR, Sabatino A, Miller S, Hanna E, Bodfish JW, Dichter GS. Common and distinct neural features of social and non-social reward processing in autism and social anxiety disorder. Soc Cogn Affect Neurosci. 2014 Mar;9(3):367-77. doi: 10.1093/scan/nss146. Epub 2012 Dec 7. PMID 23223206
- [Background] Spreckelmeyer KN, Krach S, Kohls G, Rademacher L, Irmak A, Konrad K, Kircher T, Grunder G. Anticipation of monetary and social reward differently activates mesolimbic brain structures in men and women. Soc Cogn Affect Neurosci. 2009 Jun;4(2):158-65. doi: 10.1093/scan/nsn051. Epub 2009 Jan 27. PMID 19174537
- [Background] Van Bockstaele B, Verschuere B, Tibboel H, De Houwer J, Crombez G, Koster EH. A review of current evidence for the causal impact of attentional bias on fear and anxiety. Psychol Bull. 2014 May;140(3):682-721. doi: 10.1037/a0034834. Epub 2013 Nov 4. PMID 24188418